CLINICAL TRIAL: NCT01450956
Title: The Protective Effects of Sevoflurane Application During CPB on Pediatric Patients Underwent Cardiac Surgery: a Randomized, Controlled, Blinded Clinical Trial
Brief Title: The Protective Effects of Sevoflurane in Pediatric Cardiac Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: XJXZ2011-010
Record Dates: First submitted 2011-10-07; First posted 2011-10-13 (Estimated); Last update posted 2011-11-28 (Estimated); Status verified 2011-11

CONDITIONS: Congenital Heart Diseases
Keywords: congenital heart diseases; cardiopulmonary bypass; Pediatric; sevoflurane
MeSH Terms: conditions — Heart Defects, Congenital | interventions — Sevoflurane

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sevoflurane (Experimental): Patients will receive 2% sevoflurane via oxygenator during CPB
  Interventions: Drug: Sevoflurane
- Control (No Intervention): Patients will receive only oxygen and air through oxygenator
  Interventions: Other: Control

INTERVENTIONS:
Drug: Sevoflurane — Sevoflurane will be given at a concentration of 2% through oxygenator during CPB
  Arms: Sevoflurane
Other: Control — Patients will receive only oxygen and air through oxygenator
  Arms: Control

SUMMARY:
During repair of a congenital heart defect the child is exposed to myocardial hypoxia. Recent studies have suggested that the paediatric myocardium is more sensitive to hypoxia and cardioplegic arrest than the adult. The protective effect of halogenated agents on ischaemia and reperfusion injury has been investigated widely in adults. The investigators hypothesis that sevoflurane applied during cardiopulmonary bypass might afford better myocardial protection during paediatric cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* pediatric patients (body weight < 10 kg)
* diagnosed with congenital heart diseases
* scheduled for repair operation with CPB
* in the Department of Cardiovascular Surgery, Xijing Hospital

Exclusion Criteria:

* systemic infections
* other systemic diseases

Ages: 1 Month to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2011-09; Primary Completion 2012-01 (Estimated); Study Completion 2012-01 (Estimated)

PRIMARY OUTCOMES:
all cause mortality | within the first 30 days (plus or minus 3 days) after surgery
  All cause mortality after the cardaic surgery, patients will be followed up for 30 days

SECONDARY OUTCOMES:
serum cTnI concentrations | 48 h after the surgery
  serial serum cTnI concentrations will be determined to whether sevoflurane application during CPB will decrease the cTnI release after operation.

CONTACTS AND LOCATIONS:
Overall Officials: Zhenxiao Jin, PhD, Principal Investigator — Department of Cardiovascular Surgery, Xijing Hospital
Locations (1):
- Department of Cardiovascular Surgery, Xijing Hospital, Xi'an, Shaanxi, China

REFERENCES:
- [Derived] Xiong HY, Liu Y, Shu DC, Zhang SL, Qian X, Duan WX, Cheng L, Yu SQ, Jin ZX. Effects of Sevoflurane Inhalation During Cardiopulmonary Bypass on Pediatric Patients: A Randomized Controlled Clinical Trial. ASAIO J. 2016 Jan-Feb;62(1):63-8. doi: 10.1097/MAT.0000000000000285. PMID 26418205